CLINICAL TRIAL: NCT06891131
Title: Implementation of an Empiric Transfusion Bundle for Out of Hospital Patients With Haemorrhagic Shock: a Prospective Observational Study C-TOP - Coagulation Therapy for Out-of-Hospital Patients
Brief Title: Implementation of an Empiric Transfusion Bundle for Out of Hospital Patients With Haemorrhagic Shock
Acronym: C-TOP
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1032/2025
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Haemorrhagic Shock; Trauma Coagulopathy
Keywords: Trauma; coagulopathy; haemmorhage; transfusion
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The investigators will evaluate the implementation of a treatment bundle (Fibrinogen, Plasma and Tranexamic Acid)

DETAILED DESCRIPTION:
The investigators will perform a prospective observational study of patients in haemorrhagic shock with suspected life threatening bleeding from trauma, treated by the prehospital emergency doctor response team of the Medical University of Graz and the HEMS (Helicopter Emergency Medical Service) of Graz according to their SOPs. Only patients that are being transported to the resuscitation room of the Medical University of Graz after prehospital transfusion will be included.

The SOPs for prehospital transfusion are being implemented for the treatment of patients in extremis because of suspected life-threatening traumatic bleeding in the above-mentioned emergency services, according to the manufacturer's requirements. These transfusion SOPs are already part of the standard of care in the resuscitation room of the Medical University of Graz.

This study seeks to gather information on the benefits and potential harms of this change of prehospital clinical routine.

The treatment bundle will include 2 units of Fibrinogen and Plasma in addition to 10-20 mg/kg Tranexamic Acid

ELIGIBILITY:
Inclusion Criteria:

* aged, or believed to be aged
* 18 years or above
* confirmed or suspected life-threatening bleeding from trauma (i.e. signs of inadequate perfusion of tissues, tachycardia, hypotension, suspected blood loss)
* need for volume replacement therapy.

Exclusion Criteria:

* patient with known recent history of thromboembolic events within the last 6 months
* known or suspected pregnancy at presentation
* patient with known refusal of a participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in haemorrhagic shock that are being treated by one of the prehospital emergency systems of the Medical University of Graz (HEMS, emergency car)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful prehospital bundle transfusion | prehospital setting
  to assess feasibility

SECONDARY OUTCOMES:
30-day-mortality | 30 days
blood product used in the first 24 hours | 24 hours
concentration of lactat acid ad admission | 2 hours
  measured in the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Honnef, MD, PhD, Principal Investigator — Medical University of Graz, Department of Anaesthesiology
Locations (1):
- Medical University of Graz, Graz, Austria